CLINICAL TRIAL: NCT01582529
Title: The Impact of Family Factors on Developmental and Psychosocial Outcomes in Children With Hypoplastic Left Heart Syndrome (HLHS) at 6 Years of Age - Pediatric Heart Network Single Ventricle Reconstruction Extension (SVR II) Ancillary Study
Brief Title: SVRII Family Factors Study
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Pediatric Heart Network (Other)
Responsible Party: Sponsor
Other Study IDs: 319498; U01HL068270 (NIH)
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Hypoplastic Left Heart Syndrome
Keywords: Developmental Outcomes; Psychosocial Outcomes; Hypoplastic Left Heart Syndrome; Congenital Heart Disease
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to learn about the relationship between family factors and developmental and psychosocial outcomes in children with congenital heart disease at 6 years of age. A secondary purpose is to learn more about psychosocial outcomes in children with congenital heart disease and their families over time.

About 250 mothers and fathers at 15 medical centers will take part in this study; 35 will be from Children's Hospital of Wisconsin.

DETAILED DESCRIPTION:
Survival for one of the most complex forms of congenital heart disease (CHD), hypoplastic left heart syndrome (HLHS), has improved dramatically; however, survivors are known to be at risk for both physical and psychosocial morbidity. In congenital heart disease, this psychosocial morbidity has been manifested as delays in cognitive and social development, behavior problems, reduced quality of life, as well as parenting stress, anxiety, and negative impact on the family. We have a relatively limited understanding of the causes of psychosocial morbidity and what factors may impact risk or protection for the child and family.

The environment in which a child spends the majority of their time exerts a significant impact on development. For infants and young children this "environment" is most commonly the immediate family. Interactions between illness characteristics and individual family member perceptions and expectations are an important determinant of the family's response to the presence of heart disease in a child. There is a critical gap in our understanding of how family-related factors influence psychosocial outcomes in the CHD population and if there are opportunities to intervene in order to improve outcomes for both children and families.

The primary aim of this study is to investigate the relationship between family factors including, parental mental health, parental health-related quality of life (HRQOL), family resources, and family function, and developmental and psychosocial outcomes in children with HLHS at 6 years of age. Secondary aims are to explore for differences in outcomes between different family types and to establish the feasibility of longitudinal investigation of the trajectory of child and family psychosocial function over time in this well-defined cohort of children and parents.

Longitudinal assessment of these family factors, in conjunction with neurodevelopmental and psychosocial evaluation of affected children, will provide improved understanding of how and when these factors influence child development. This will help to:

* Identify children/families at risk for problems,
* Elucidate the etiology and progression of psychosocial problems in children with congenital heart disease,
* Describe the relationships between child and family outcomes over time, and guide the development of family-focused interventions with a goal of preventing problems.

This study will be conducted as an ancillary study to the Single Ventricle Reconstruction Extension Study (SVR II) conducted by the Pediatric Heart Network (PHN). All PHN study sites will be eligible to participate in this study. Participation will be determined by the PHN principal investigator at each site. Parents of children enrolled in SVR II will be eligible to participate in this ancillary study.

A multivariable, descriptive design using survey techniques will be utilized. Mothers and fathers of children with HLHS will complete study measures at or near the SVR II 6 year visit. Correlation, regression, and structural equation modeling will be used to test study hypotheses.

Results of this study have the potential to better define the family implications of this disease, the risk factors for poor outcomes and ultimately, to guide development of interventions to improve child and family psychosocial outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Speak English or Spanish
* Enrolled in the SVR or SVRII studies

Exclusion Criteria:

* Have not completed the 6 year visit and questionnaires

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Parents of subjects that are enrolled in the "Single Ventricle Reconstructive Extension Study" (SVR) or the SVR II study sponsored by the Pediatric Heart Network.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
Parental mental health | During child's 6th year of life.
  Parental mental health will be assessed with the Patient-Reported Outcomes Measurement Information System (PROMIS) anxiety and depression scales.
Parental quality of life | During child's 6th year of life.
  Parental quality of life will be assessed with the Satisfaction with Health and Life Scale (SHL) (also referred to as the Perceived Quality of Life Scale).
Family resources | During child's 6th year of life
  Family resources will be assessed with the Family Inventory of Resources for Management (FIRM.
Family function | During child's 6th year of life
  Family function will be assessed with the Family Assessment Device (FAD)39 and the Family Management Measure (FaMM.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Mussatto, PhD, RN, Principal Investigator — Children's Hospital and Health System Foundation, Wisconsin
Locations (11):
- United States (10):
  - Children's Hospiral of Los Angeles, Los Angeles, California
  - Nemours/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Hospital Boston, Boston, Massachusetts
  - The University of Michigan, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- The Hospital for Sick Children, Toronto, Ontario, Canada